CLINICAL TRIAL: NCT05479500
Title: Investigation of the Efficacy of Myofascial Chain Release Techniques on Plantar Fasciitis Pain, Lower Extremity Functional Capacity and Quality of Life - Randomized Controlled Study
Brief Title: Investigation of the Efficacy of Myofascial Chain Release Techniques on Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ayca Evkaya Acar, Lecturer, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/0346
Record Dates: First submitted 2022-07-22; First posted 2022-07-29 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Plantar Fascitis
Keywords: Plantar Fascitis; Fascia; Myofascial Release Techniques

STUDY DESIGN:
Intervention Model Description: There will be three groups in this study. Each group will consist of 12 patients aged 30-60 years with plantar fasciitis. A total of 36 participants will take part in the study. Conventional physiotherapy will be applied to the group 1 and, local release technique addition to conventional physiotherapy will be applied to the group 2, while myofascial release techniques will be applied to the experimental group in addition to conventional physiotherapy.
Who Masked: Outcomes Assessor
Masking Description: Participants will be divided into three groups using block randomization method. Participants will be randomly allocated into 3 blocks of 12 participants in each group using a random number generation technique by computer. All assessments will be done by researcher who were not in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (No Intervention): Control group will consist of 12 patients with diagnosed Plantar Fasciitis, aged between 30-60 years. Only conventional physiotherapy program will be applied to this group.
  Conventional treatment will consist of foot intrinsic muscles strengthening, plantar fascia, achilles and hamstring stretching exercises. The exercises will be performed as 10 repetitions and 3 sets. Participants will be treated for a total of 6 weeks, 2 days a week. Each treatment session will last 20-40 minutes.
- Group 2 (Experimental): Experimental group will consist of 12 patients with diagnosed Plantar Fasciitis, aged between 30-60 years. In addition to the conventional physiotherapy program, local release techniques will be applied to this group. Local Release Techniques will be applied as Gastro-solues trigger point myofascial release and Plantar fascia myofascial release. Participants will be treated for a total of 6 weeks, 2 days a week. Each treatment session will last 20-40 minutes.
  Interventions: Other: Local Release Techniques
- Group 3 (Experimental): Experimental group will consist of 12 patients with diagnosed Plantar Fasciitis, aged between 30-60 years. In addition to the conventional physiotherapy program, myofascial chain release techniques will be applied to this group.
  Myofascial release technique will be applied to the center of coordination points in the superficial back line myofascial chain of the body. Pressure will be applied to each point with 6 repetitions and lasting approximately 5-6 seconds.
  Participants will be treated for a total of 6 weeks, 2 days a week. Each treatment session will last 20-40 minutes.
  Interventions: Other: Myofascial Chain Release Techniques

INTERVENTIONS:
Other: Myofascial Chain Release Techniques — Myofascial release is a hands on technique which stretches the fascia and releases, bonds between muscles, integuments and fascia in order to eliminate pain, improve motion and to maintain myofascial balance within the body.
  Arms: Group 3
Other: Local Release Techniques — Local Release Techniques are a soft tissue method that focuses on relieving tissue tension via the removal of fibrosis/adhesions which can develop in tissues as a result of overload due to repetitive use.
  Arms: Group 2

SUMMARY:
The primary aim of the study is to investigate the effectiveness of Myofascial Chain Release Techniques on pain, functional limitation and quality of life in patients with Plantar Fasciitis. The secondary aim of the study is to create a future clinical projection regarding the applications to be made over the myofascial chain in addition to the generally accepted treatment protocols in the light of the findings.

There will be three groups in this study. Each group will consist of 12 patients aged 30-60 years with plantar fasciitis. A total of 36 participants will take part in the study. Conventional physiotherapy will be applied to the group 1 and, local release technique addition to conventional physiotherapy will be applied to the group 2, while myofascial release techniques will be applied to the experimental group in addition to conventional physiotherapy. Treatment programs will be applied to both groups 2 days a week for 6 weeks. Postural problems that can be seen in the superficial back myofascial chain line will be evaluated.

DETAILED DESCRIPTION:
The plantar fascia is an important connective structure that extends from the metatarsal heads to the calcaneus and provides the continuity of the longitudinal arch of the foot. Microtraumas and the formation of chronic inflammation on the plantar surface, which is exposed to repetitive stress, thickens the fascia, making it susceptible to repetitive injuries and forming plantar fasciitis. The reasons for this repetitive stress are; excessive physical activity, obesity, age, prolonged standing, biomechanical changes, limited dorsiflexion and hamstring tension.

Studies on this subject in the literature have reported that tension in the hind leg muscles is associated with plantar fasciitis, and applications on the Achilles tendon and gastrocnemius have been shown to relieve plantar fasciitis complaints. Similarly, it has been reported that tension in the hamstring muscle may be associated with the development of plantar fasciitis.

It is known that the Plantar Fascia and Achilles tendon affect each other due to the fascial connection, and therefore these structures are considered together in the solution of their problems. On the other hand, according to the fascial meridian concept developed by Thomas Myers, it was stated that the fascial connection between these two tissues extends to the frontal region in a chain manner, and that a problem at any point in the chain may cause problems in other elements of the chain. For this reason, recently, applications related to the detection and solution of problems have come to the fore by looking at fascial problems more holistically over the fascial chain. From this point of view, there are many studies reporting the effectiveness of applications performed in any region of the myofascial chain in a different region on this chain.

Plantar Fascia; It is located in the Superficial Back Line, and as far as we know, there is no study of plantar fasciitis treatment in which the myofascial chain is considered as a whole. Based on this, our aim in this study is to investigate the effect of myofascial release techniques applied along the myofascial chain line on pain, lower extremity functionality and quality of life in patients diagnosed with Plantar fasciitis. In the light of the findings, it is to create a projection for future clinical studies regarding the treatment approaches to be applied over the myofascial chain in addition to the generally accepted treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between the ages of 30-60
* Diagnosed with plantar fasciitis
* Not having received medical treatment and/or physiotherapy for plantar fasciitis in the last 3 months.
* The participants' definition of pain over 3 according to the Visual Analogue Scale in the first step of the morning and this pain decreases with movements

Exclusion Criteria:

* Having history of lower extremity surgery and fracture in the last 6 months
* Having additional orthopedic, neurological and rheumatological diseases that may cause biomechanical malalignment, loss of muscle strength, and deterioration of gait parameters in the lower extremities, vertebral column and pelvis
* Having static foot deformity
* Having connective tissue disease that will affect tissue properties
* Having metabolic syndromes that may affect tissue properties such as diabetes
* Using sedatives and/or muscle relaxants that may alter muscle tone.
* Being diagnosed with obesity (BMI>30)
* Pregnancy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Ultrasonography | Change from baseline ultrasonography at week 6.
  It will be used to measure the thickness of the plantar fascia. As a result of these studies, a plantar fascia greater than 4 mm appears to be abnormal and associated with plantar fasciitis. Ultrasonography (USG) evaluation is a routine method for the diagnosis of Plantar Fasciitis.
Plantar Fasciitis Pain | Change from baseline plantar fasciitis pain at week 6.
  Visual Analogue Scale will be used in the assessment of pain severity. It expresses pain severity between a score of 0 (no pain) and 10 (unbearably severe pain).
Pes planus | Change from baseline pes planus at week 6.
  Pes Planus will be evaluated with navicular drop test. The distance between the navicular bone and the ground is measured while the individual sits on the chair with the hip-knee joint in 90º flexion and the subtalar joint in neutral position. Then, the distance between the navicular bone and the ground is measured again while the individual is standing in a position with equal weight on both extremities. The difference between the two measurements is recorded. 10 mm or more difference is considered pes planus.
Foot Posture | Change from baseline foot posture at week 6.
  Foot posture will be evaluated using the Foot posture index, a six item foot posture assessment tool, where each item is scored between -2 and +2 to give a sum total between -12 (highly supinated) and +12 (highly pronated). Items include: talar head palpation, curves above and below the lateral malleoli, calcaneal angle, talonavicular bulge, medial longitudinal arch, and forefoot to rearfoot alignment.
Ankle Joint Angle | Change from baseline ankle joint angles at week 6.
  Active and passive dorsi and plantar flexion angles will be measured with a goniometer.
Algometer | Change from baseline pressure pain threshold at week 6.
  It is used to measure the pressure pain threshold. After localization of the painful area by palpation, force is applied with an algometer until patients feel pain and discomfort. The digit displayed on the algometer is recorded. The average of 3 measurements is taken.
Passive Tone | Change from baseline passive tone of myofascial tissues at week 6.
  Passive Tone will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Stiffness | Change from baseline Stiffness of myofascial tissues at week 6.
  Stiffness will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Decrement | Change from baseline Decrement of myofascial tissues at week 6.
  Decrement will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Creep | Change from baseline Creep of myofascial tissues at week 6.
  Creep will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Relaxation time | Change from baseline Relaxation time of myofascial tissues at week 6.
  Relaxation time will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Hamstring Muscle shortness | Change from baseline Hamstring muscle shortness at week 6.
  Hamstring length will be measured with the straight leg lift test. The patient is asked to keep the opposite leg fixed on the bed with the knee straight in the supine position, wearing suitable clothes, and to raise the leg to be tested upwards with the ankle in dorsiflexion and the knee straight. The patient is instructed to wait where the initial tension occurs, and the last degree of movement is measured.
Pelvic tilt | Change from baseline pelvic tilt at week 6.
  The position of the pelvis will be evaluated with a digital pelvic inclinometer device to determine whether the pelvis has tilted anteriorly or posteriorly. The digital pelvic inclinometer is a valid and reliable method for the evaluation of pelvic tilt. The device consists of two calipers and the calipers are placed on the spina iliaca anterior superior (SIAS) and spina iliaca posterior superior (SIPS) of the pelvis. The score on the digital display is recorded. "-" values indicate posterior pelvic tilt, "+" values indicate anterior pelvic tilt.
Cervical and Lumbar Lordosis | Change from baseline Cervical and Lumbar Lordosis at week 6.
  It will be determined by photographing. Side photos will be taken while the patient is standing in a free standing position in front of a bare, flat wall with the upper body. Later, the obtained photo shoots will be analyzed with the Tracker 4.11.0 (Physlets, 2017) program and cervical and lumbar lordosis angles will be determined.
Skin temperature of the Plantar Fascitis area | Change from baseline Skin temperature of the Plantar Fascitis area at week 6.
  In order to see the effectiveness of the applications, the skin temperature will be determined by thermal imaging method. This method is frequently preferred because it is a reliable and non-invasive method. The skin temperature of the plantar fascia will be measured with the P45 thermographic camera (Flir System, ThermaCAM, Sweden) with high thermal sensitivity, while the patient is in the prone position, while the feet are hanging from the bed at the level of the malleolus. The measurement will be made by placing the camera on a tripod placed 1m away from the patient. In the analysis, the area covering 1 cm distance from the point where fasciitis develops will be used. Skin temperature will be determined using the FLIR Quick-Report 1.2 software, one of the temperature indicators obtained from this region. In the calculation of skin temperature, the human skin emissivity value will be accepted as 0.98.
Headache | Change from baseline Headache at week 6.
  Presence of headache will be questioned and severity assessment will be made with Visual Analogue Scale. It expresses pain severity between a score of 0 (no pain) and 10 (unbearably severe pain).
Windlass Test | Change from baseline Windlass Test at week 6.
  While the patient is sitting in a chair, the big toe of the foot to be tested is brought into the dorsal flexion of the metatarsal phalangeal joint for a hard time. Pain at the junction of the plantar fascia with the calcaneus during this movement indicates a positive test.
SF-12 Quality of Life | Change from baseline Quality of Life at week 6.
  An abbreviated form for assessing quality of life. SF-12, a form developed in 1994, is not specific to any age and disease type, and is a scale that evaluates the quality of life of the person during the last four weeks. SF-12; physical functionality includes physical role, pain, general health, emotional role, mental health, social functionality and vitality.
Lower extremity functionality | Change from baseline lower extremity functionality at week 6.
  Lower extremity functional scale will be used. This scale is a valid and reliable scale used in musculoskeletal problems affecting the lower extremities. It consists of 20 items. Each item is scored between 0-4. The total score is between 0-80. Higher scores indicate better functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Kablan, Asst. Prof., Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JH, Jung HW, Jang WY. A prospective study of the muscle strength and reaction time of the quadriceps, hamstring, and gastrocnemius muscles in patients with plantar fasciitis. BMC Musculoskelet Disord. 2020 Nov 5;21(1):722. doi: 10.1186/s12891-020-03740-1. PMID 33153452
- [Background] Williams W, Selkow NM. Self-Myofascial Release of the Superficial Back Line Improves Sit-and-Reach Distance. J Sport Rehabil. 2019 Oct 18;29(4):400-404. doi: 10.1123/jsr.2018-0306. Print 2020 May 1. PMID 30860410
- [Background] Burk C, Perry J, Lis S, Dischiavi S, Bleakley C. Can Myofascial Interventions Have a Remote Effect on ROM? A Systematic Review and Meta-Analysis. J Sport Rehabil. 2019 Oct 18;29(5):650-656. doi: 10.1123/jsr.2019-0074. Print 2020 Jul 1. PMID 31629335
- [Background] Arshad Z, Aslam A, Razzaq MA, Bhatia M. Gastrocnemius Release in the Management of Chronic Plantar Fasciitis: A Systematic Review. Foot Ankle Int. 2022 Apr;43(4):568-575. doi: 10.1177/10711007211052290. Epub 2021 Nov 12. PMID 34766860
- [Background] Hoefnagels EM, Weerheijm L, Witteveen AG, Louwerens JK, Keijsers N. The effect of lengthening the gastrocnemius muscle in chronic therapy resistant plantar fasciitis. Foot Ankle Surg. 2021 Jul;27(5):543-549. doi: 10.1016/j.fas.2020.07.003. Epub 2020 Jul 12. PMID 32773360
- [Background] Martinez-Lema D, Guede-Rojas F, Gonzalez-Fernandez K, Soto-Martinez A, Lagos-Hausheer L, Vergara-Rios C, Marquez-Mayorga H, Mancilla CS. Immediate effects of a direct myofascial release technique on hip and cervical flexibility in inactive females with hamstring shortening: A randomized controlled trial. J Bodyw Mov Ther. 2021 Apr;26:57-63. doi: 10.1016/j.jbmt.2020.12.013. Epub 2020 Dec 11. PMID 33992297
- [Background] Dhiman NR, Das B, Mohanty C, Singh OP, Gyanpuri V, Raj D. Myofascial release versus other soft tissue release techniques along superficial back line structures for improving flexibility in asymptomatic adults: A systematic review with meta-analysis. J Bodyw Mov Ther. 2021 Oct;28:450-457. doi: 10.1016/j.jbmt.2021.06.026. Epub 2021 Jun 16. PMID 34776177
- [Background] Fauris P, Lopez-de-Celis C, Canet-Vintro M, Martin JC, Llurda-Almuzara L, Rodriguez-Sanz J, Labata-Lezaun N, Simon M, Perez-Bellmunt A. Does Self-Myofascial Release Cause a Remote Hamstring Stretching Effect Based on Myofascial Chains? A Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Nov 24;18(23):12356. doi: 10.3390/ijerph182312356. PMID 34886078